CLINICAL TRIAL: NCT06856447
Title: The Role of Coenzyme Q10 in the Prophylaxis of Oxaliplatin Induced Peripheral Neuropathy in Patients With Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: toqa saad mohammed mohammed (Other)
Responsible Party: Sponsor-Investigator, toqa saad mohammed mohammed, Master's Researcher in Clinical Pharmacy, Tanta University, Tanta University
Organization: Tanta University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Prophylaxis of neuropathy
Record Dates: First submitted 2024-06-03; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer
Keywords: Oxaliplatin-induced neuropathy; Coenzyme Q10; Neuroprotection in cancer; Chemotherapy-induced neuropathy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — coenzyme Q10; Oxaliplatin; Fluorouracil; Serotonin 5-HT3 Receptor Antagonists; Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control group (Placebo Comparator): Patients in the control group will receive 12 cycles of the modified FOLFOX-6 regimen, which consists of oxaliplatin, 5-fluorouracil (5-FU), and leucovorin, administered every two weeks. Supportive care includes an intravenous 5-HT3 antagonist for nausea prevention and pantoprazole to prevent gastric irritation.
  Interventions: Drug: Oxaliplatin; Drug: 5-Fluorouracil (5-FU); Drug: 5-HT3 Antagonist; Drug: Pantoprazole
- Experimental (Experimental): Patients in the experimental group will receive 12 cycles of the modified FOLFOX-6 regimen with the same supportive medications as the control group. Additionally, they will receive Coenzyme Q10 (100 mg once daily in the morning), starting after the first chemotherapy cycle and continuing until the end of the 12th cycle.
  Interventions: Drug: Coenzyme Q10; Drug: Oxaliplatin; Drug: 5-Fluorouracil (5-FU); Drug: 5-HT3 Antagonist; Drug: Pantoprazole

INTERVENTIONS:
Drug: Coenzyme Q10 — 100 mg once daily starting after the first chemotherapy cycle. Patients will receive 12 cycles of the modified FOLFOX-6 regimen with Coenzyme Q10 (100 mg once daily in the morning), starting after the first chemotherapy cycle and continuing until the end of the 12th cycle. Based on McRae (2023), 200 mg/day for 12 weeks reduced TNF-α and IL-6; thus, 100 mg/day for 6 months was selected (one cycle every 2 weeks = 24 weeks).
  Supportive care: Includes a 5-HT3 antagonist for nausea prevention and pantoprazole to prevent gastric irritation.
  Intervention Details:
  Oxaliplatin: Part of the FOLFOX-6 regimen. 5-Fluorouracil (5-FU): Part of the FOLFOX-6 regimen. Leucovorin: Part of the FOLFOX-6 regimen. 5-HT3 Antagonist: Used for nausea prevention. Pantoprazole: Used to prevent gastric irritation.
  Other Names: Coenzyme Q10 Forte
  Arms: Experimental
Drug: Oxaliplatin — Part of the modified FOLFOX-6 chemotherapy regimen
Drug: 5-Fluorouracil (5-FU) — Part of the modified FOLFOX-6 chemotherapy regimen.
Drug: 5-HT3 Antagonist — Used for nausea prevention during chemotherapy.
Drug: Pantoprazole — Used to prevent gastric irritation during chemotherapy

SUMMARY:
This study aims to evaluate the possible beneficial role of coenzyme Q10 against oxaliplatin-induced peripheral neuropathy in patients with colorectal cancer.

DETAILED DESCRIPTION:
Oxaliplatin (OXA), a third-generation platinum-based anticancer drug, has better efficacy and lower toxicity than cisplatin and carboplatin. Currently, OXA combined with 5-FU and leucovorin is the standard adjuvant chemotherapy regimen for colorectal cancer (CRC) and the first-line treatment for metastatic CRCs. The major side effects of OXA include peripheral neurotoxicity, myelosuppression, and diarrhea. These adverse effects may lead to treatment discontinuation and reduced compliance among CRC patients. Specifically, oxaliplatin-induced peripheral neuropathy (OIPN) is a dose-limiting toxicity associated with OXA.

The mechanisms involved in OIPN include functional abnormalities in voltage-gated K+ channels, with increased expression of pro-excitatory K+ channels such as hyperpolarization-activated channels. Abnormalities in Na+ currents have been detected in 78% of patients who later develop chronic OXA-induced neuropathy (Krishnan et al., 2005). Dysregulation of Ca2+ homeostasis has also been suggested as a key factor in OXA-associated nerve damage. In vivo studies indicate that oxaliplatin-induced cold allodynia enhances the sensitivity and expression of transient receptor potential A1 (TRPA1) and transient receptor potential cation channel subfamily M member 8 (TRPM8).

Several studies suggest a relationship between OXA-induced neuropathy and oxidative stress. Additional potential contributors to neuropathic pain include T-cells (Th17 and Th1) and inflammatory cytokines such as tumor necrosis factor-alpha (TNF-α). Clinical studies have demonstrated that elevated IL-6 levels correlate with painful chemotherapy-induced neuropathy, and patients receiving IL-6 neutralizing antibodies as part of their therapy report reduced neuropathic pain compared to those not receiving these antibodies.

Coenzyme Q10 (CoQ10) is an oil-soluble, vitamin-like substance primarily present in mitochondria. It possesses anti-inflammatory and antioxidant properties and has demonstrated neuroprotective effects in animal models of neurodegeneration by stimulating cell growth and inhibiting cell death. CoQ10 has been shown to protect against cisplatin-induced neurotoxicity in a rat model and to reduce paclitaxel-induced peripheral neuropathy in rodents. Additionally, CoQ10 exhibited a protective effect against vincristine-induced peripheral neuropathy in rats (Elshamy et al., 2022). The neuroprotective effects of CoQ10 have been attributed to its ability to mitigate oxidative stress and inflammation, evidenced by significant reductions in malondialdehyde (MDA), 8-hydroxyguanosine (8-OHdG), TNF-α, IL-1β, and nuclear factor kappa-B. CoQ10 has also been reported to lower serum neurofilament-light chain (NF-L), a recognized biomarker for multiple neurodegenerative diseases.

In diabetic patients with peripheral neuropathy, antioxidant and anti-inflammatory supplementation with CoQ10 has shown potential benefits. A study reported that administration of CoQ10 at a dose of 200 mg/day for 12 weeks in neuropathic diabetic patients improved total antioxidant capacity (TAC) and reduced high-sensitivity C-reactive protein (hsCRP).

To the best of the investigators' knowledge, no clinical trials have been conducted to evaluate CoQ10 as a prophylactic therapy against chemotherapy-induced neuropathy. This study aims to assess its potential role in preventing oxaliplatin-induced peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosis of Stage III colorectal cancer.
* Patients who will be scheduled to receive modified FOLFOX-6.
* Patients with no contraindication to chemotherapy.
* Males and females aged ≥ 18 years old.
* Adequate baseline hematologic values (absolute neutrophilic count ≥ 1.5 × 109 /L, platelet count ≥ 100 × 109 /L and hemoglobin level ≥ 10 g/dl).
* Patients with adequate renal function (serum creatinine < 1.5 mg/dl
* Patients with adequate liver function (serum bilirubin < 1.2 mg/dl).
* Patients with performance status 0-1 according to Eastern Cooperative Oncology Group (ECOG) score.
* Patients who may receive medications to counteract chemotherapy induced neuropathic pain (gabapentin, lamotrigine, carbamazepine, etc….).

Exclusion Criteria:

* Exclusion criteria

  * Patients with prior exposure to neurotoxic agents (Cisplatin, vincristine, paclitaxel, docetaxol, foscarnet, INH, etc..) in the last 6 months.
  * Patients with evidence of metastasis at the initial assessment.
  * Concomitant use of antioxidant vitamins (vitamin A, C, E),
  * Preexisting peripheral neuropathy resulting from other causes such as diabetes and brain disorders, hypothyroidism, autoimmune diseases, hepatitis C.
  * Patients with diabetes.
  * Patients with inflammatory diseases (ulcerative colitis, rheumatoid arthritis).
  * Patients with stressful conditions as smoking, COPD, ….
  * Patients with active liver disease (cirrhosis, fatty liver, hepatitis C, etc..).
  * Patients with myopathy
  * Patients with renal impairment, including those with end-stage renal disease and those receiving dialysis.
  * Pregnant and breast feeding women.
  * Concurrent use of diltiazem, metoprolol, enalapril, nitroglycerin, warfarin, clopidigrel, aspirin, statins, fibrates, tricyclic antidepressant medications,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Tumor necrosis factor-alpha (TNF-α) | Between 8:30 AM and 10:30 AM after overnight fasting. Blood samples will be collected into a plain test tube and centrifuged at 3,000 revolutions per minute (RPM) for 10 minutes.
  Tumour Necrosis Factor alpha (TNF alpha), is an inflammatory cytokine produced by macrophages/monocytes during acute inflammation and is responsible for a diverse range of signalling events within cells, leading to necrosis or apoptosis.

SECONDARY OUTCOMES:
Neurofilament-light chain (NF-L). | Between 8:30 AM and 10:30 AM after overnight fasting. Blood samples will be collected into a plain test tube and centrifuged at 3,000 revolutions per minute (RPM) for 10 minutes.
  eurofilament-light chain (Nf-L) is a reliable biomarker in the context of neurodegenerative diseases (NDD) and traumatic brain injuries (TBI).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Reda Kelany, dr, Study Director — Associate Professor of Clinical Oncology Faculty of Medicine - Ain-Shams University; Eman Ibrahim Abd Elkader Elberri, Study Director — Lecturer of Clinical Pharmacy Faculty of Pharmacy - Tanta University
Locations (1):
- Ain-Shams University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kidwell KM, Yothers G, Ganz PA, Land SR, Ko CY, Cecchini RS, Kopec JA, Wolmark N. Long-term neurotoxicity effects of oxaliplatin added to fluorouracil and leucovorin as adjuvant therapy for colon cancer: results from National Surgical Adjuvant Breast and Bowel Project trials C-07 and LTS-01. Cancer. 2012 Nov 15;118(22):5614-22. doi: 10.1002/cncr.27593. Epub 2012 May 8. PMID 22569841
- [Background] Krishnan AV, Goldstein D, Friedlander M, Kiernan MC. Oxaliplatin-induced neurotoxicity and the development of neuropathy. Muscle Nerve. 2005 Jul;32(1):51-60. doi: 10.1002/mus.20340. PMID 15880395
- [Background] Marmiroli P, Riva B, Pozzi E, Ballarini E, Lim D, Chiorazzi A, Meregalli C, Distasi C, Renn CL, Semperboni S, Morosi L, Ruffinatti FA, Zucchetti M, Dorsey SG, Cavaletti G, Genazzani A, Carozzi VA. Susceptibility of different mouse strains to oxaliplatin peripheral neurotoxicity: Phenotypic and genotypic insights. PLoS One. 2017 Oct 11;12(10):e0186250. doi: 10.1371/journal.pone.0186250. eCollection 2017. PMID 29020118
- [Background] McRae MP. Coenzyme Q10 Supplementation in Reducing Inflammation: An Umbrella Review. J Chiropr Med. 2023 Jun;22(2):131-137. doi: 10.1016/j.jcm.2022.07.001. Epub 2022 Aug 31. PMID 37346240
- [Background] Nassini R, Gees M, Harrison S, De Siena G, Materazzi S, Moretto N, Failli P, Preti D, Marchetti N, Cavazzini A, Mancini F, Pedretti P, Nilius B, Patacchini R, Geppetti P. Oxaliplatin elicits mechanical and cold allodynia in rodents via TRPA1 receptor stimulation. Pain. 2011 Jul;152(7):1621-1631. doi: 10.1016/j.pain.2011.02.051. Epub 2011 Apr 9. PMID 21481532
- [Background] Nielsen DL, Palshof JA, Larsen FO, Jensen BV, Pfeiffer P. A systematic review of salvage therapy to patients with metastatic colorectal cancer previously treated with fluorouracil, oxaliplatin and irinotecan +/- targeted therapy. Cancer Treat Rev. 2014 Jul;40(6):701-15. doi: 10.1016/j.ctrv.2014.02.006. Epub 2014 Feb 28. PMID 24731471
- [Background] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Background] Sommer C, Kress M. Recent findings on how proinflammatory cytokines cause pain: peripheral mechanisms in inflammatory and neuropathic hyperalgesia. Neurosci Lett. 2004 May 6;361(1-3):184-7. doi: 10.1016/j.neulet.2003.12.007. PMID 15135924
- [Background] Tan G, Jensen MP, Thornby JI, Shanti BF. Validation of the Brief Pain Inventory for chronic nonmalignant pain. J Pain. 2004 Mar;5(2):133-7. doi: 10.1016/j.jpain.2003.12.005. PMID 15042521